CLINICAL TRIAL: NCT06237231
Title: Phase III, Multicenter, Double-blind, Triple-dummy, Randomized, Parallel Clinical Trial to Evaluate the Efficacy and Safety of DIT112 in the Treatment of Moderate to Severe Pain After Dental Surgery for the Extraction of Impacted Third Molars
Brief Title: Efficacy and Safety of DIT112 in the Treatment of Moderate to Severe Pain After Dental Surgery for the Extraction of Impacted Third Molars
Acronym: ALIV
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DIT112-III-0123
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Moderate Pain; Severe Pain
Keywords: pain
MeSH Terms: conditions — Pain | interventions — Dipyrone; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DIT112 (Experimental): The study is triple-dummy. The patient must take 3 pills, with a minimum interval of 6/6 hours for 3 days, if pain, as follows:
  1 tablet DIT112, oral;
  1 capsule tramadol placebo, oral;
  1 tablet dipyrone placebo, oral.
  Interventions: Drug: DIT112; Drug: Dipyrone Placebo; Drug: Tramadol Placebo
- DIPYRONE (Active Comparator): The patient must take 3 pills, with a minimum interval of 6/6 hours for 3 days, if pain, as follows:
  1 tablet dipyrone, oral;
  1 tablet DIT112 placebo, oral;
  1 capsule tramadol placebo, oral.
  Interventions: Drug: DIPYRONE; Drug: DIT112 Placebo; Drug: Tramadol Placebo
- TRAMADOL (Active Comparator): The patient must take 3 pills, with a minimum interval of 6/6 hours for 3 days, if pain, as follows:
  1 capsule tramadol, oral;
  1 tablet dipyrone placebo, oral;
  1 tablet DIT112 placebo, oral.
  Interventions: Drug: TRAMADOL; Drug: DIT112 Placebo; Drug: Dipyrone Placebo

INTERVENTIONS:
Drug: DIT112 — DIT112 tablet
  Arms: DIT112
Drug: DIPYRONE — Dipyrone tablet 1.000mg
  Arms: DIPYRONE
Drug: TRAMADOL — Tramadol tablet 50mg
  Arms: TRAMADOL
Drug: DIT112 Placebo — DIT112 placebo tablet
  Arms: DIPYRONE; TRAMADOL
Drug: Dipyrone Placebo — Dipyrone placebo tablet
  Arms: DIT112; TRAMADOL
Drug: Tramadol Placebo — Tramadol placebo capsule
  Arms: DIPYRONE; DIT112

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of DIT112 in adolescents and adults with acute pain after dental surgery for the extraction of impacted third molars.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree with all the purposes of the trial, signing and dating the Free and Informed Consent Form (TCLE) and/or the Free and Informed Assent Form (TALE) in two copies;
* Age equal to or over 15 years old;
* Indication of extraction of two (02) impacted third molars, one (01) lower third molar and one (01) upper molar on the same side;
* Third molar with bone impactions observed through panoramic radiography, with classification by Winter (1926) (1) mesioangular or vertical, and classification according to Pell & Gregory (1933) (2):

  i. Class II position B; or ii. Class III position A or B
* Presence of pain of moderate or severe intensity (score greater than or equal to 5 when assessed using an 11-point numeric pain scale) within up to four (04) hours after the end of the surgery.

Exclusion Criteria:

* Presence of local conditions (lesions in the region of the third molars) that may interfere with the extraction of third molars, such as, but not limited to, pericoronitis, periodontitis, tumors, cysts and inflammation and/or infection in the region to be operated;
* Presence of any clinical observation finding (clinical/physical assessment) or laboratory condition that is interpreted by the investigating physician as a risk to the research participant's participation in the clinical trial or the presence of uncontrolled chronic disease(s);
* Presence of a known gastroduodenal ulcer or diagnosis of persistent gastritis;
* Presence of compromised bone marrow function or diseases of the hematopoietic system;
* Presence of known severe renal and/or hepatic insufficiency;
* Diagnosis of epilepsy not adequately controlled;
* Diagnosis of acute intermittent hepatic porphyria;
* Presence of known congenital glucose-6-phosphatedehydrogenase deficiency;
* History of allergy or intolerance to tramadol, diclofenac and pyrazolones (e.g. phenazone, propyphenazone) or pyrazolidines (e.g. phenylbutazone, oxyphenbutazone) including, for example, previous experience of agranulocytosis with one of these substances;
* Use of sedative, hypnotic or psychotropic medications in the last 24 hours before surgery;
* Use of anticoagulant medications in the last seven (07) days before surgery;
* Current chronic treatment with opioids or corticosteroids;
* Current treatment with selective cyclooxygenase - 2 (COX2) inhibitors;
* Use of monoamine oxidase inhibitors (MAOIs) such as, but not limited to, phenelzine, tranylcypromine and isocarboxazid, in the last 14 days prior to the day of surgery;
* Use of any analgesic and/or anti-inflammatory medication in the three (03) days prior to the day of surgery;
* Known allergy or hypersensitivity to the components of the medicines used during the clinical trial;
* Surgery to extract third molars lasting more than 60 minutes, considering from the beginning of the incision until the end of the extraction;
* Technical failure in anesthesia or need to administer more than three tubes of anesthetic for each molar;
* Presence of temporomandibular joint dysfunction or limited mouth opening;
* Occurrence of a surgical accident resulting from the extraction of impacted third molars which, in the opinion of the investigator, could interfere with the procedures or evaluations of the trial, such as, but not limited to, intraoperative hemorrhage, probable injury to the inferior alveolar nerve, board fracture bone and soft tissue laceration;
* Current medical history of cancer and/or cancer treatment in the last 5 years;
* History of alcohol and/or illicit drug abuse disorder in the last two (02) years;
* Participants who are pregnant, breastfeeding or planning to become pregnant, or female participants of childbearing potential who are not using a reliable method of contraception;
* Participation in clinical trial protocols in the last 12 (twelve) months (CNS Resolution 251, of August 7, 1997, item III, subitem J), unless the investigator believes that there may be a direct benefit to the participant.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2027-04-10 (Estimated)

PRIMARY OUTCOMES:
Total pain relief within four (04) hours after the first PSI administration, assessed using the area under the curve of pain interruption scores (TOTPAR0-4h). | 0-4 hours
  (TOTPAR4), with pain relief assessed using a 5-point categorical scale (0 = no relief, 1 = little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief) at times 0.5, 1, 2, 3 and 4 hours.

SECONDARY OUTCOMES:
Total pain relief within six (06) hours after the first PSI administration, assessed using the area under the curve of pain interruption scores (TOTPAR0-6h). | 0-6 hours
  (TOTPAR6), with pain relief assessed using a 5-point categorical scale (0 = no relief, 1 = little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief) at times 0.5, 1, 2, 3,4, 5 and 6 hours.
Pain intensity in periods of four (04) and six (06) hours after the first PSI administration, assessed through the difference in pain intensity score (SPID0-4h and SPID0-6h, respectively). | 0-4 hours and 0-6 hours, respectively
  pain intensity four (04) hours and six (06) hours after administration of the first dose of the PSI (SPID0-4 and SPID0-6h, respectively) using an 11-point numerical scale (0 to 10 points, with 0 = absence of pain and 10 = worst possible pain) in times 0, 0.5, 1, 2, 3, 4, 5 and 6 hours.
Use of the rescue medication (time for the first use of the rescue medication within the first 24 hours after the first PSI administration); | 24 hours
  medication accounting
Overall effectiveness of the treatment according to the participant 24 hours after the first administration of the PSI (distribution of participants according to a 5-point categorical scale). | 24 hours
  Global assessment of the treatment by the participant 24 hours after administration of the first dose of PSI, using a 5-point categorical scale (0 = much worse, 1 = worse, 2 = the same, 3 = better, 4 = much better).